CLINICAL TRIAL: NCT05607875
Title: The Development and Efficacy of the Grow to Recovery Train-the-Trainer Program
Brief Title: The Grow to Recovery Train-the-Trainer Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B-ER-108-428
Record Dates: First submitted 2022-10-23; First posted 2022-11-07 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Mental Disorders; Recovery
Keywords: recovery program
MeSH Terms: conditions — Mental Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Grow to Recovery train-the-trainer group (Experimental): Professionals of the train-the-trainer group will receive an online training and then conduct a recovery group.
  Interventions: Behavioral: The Grow to Recovery Train-the-Trainer program
- Control group (Other): Professionals of the control group will not receive training.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: The Grow to Recovery Train-the-Trainer program — Mental health professionals will receive an online training, a trainer manual, a recovery manual (for people with mental illness), and "Pathways to Recovery: A Strengths Recovery Self-help Workbook". The online training includes the concept of recovery, the implementation of recovery-oriented services, and the introduction of the Grow to recovery group. After the training, these professionals will conduct a 5-month Grow to recovery group in their own organization.
  People with mental illness will attend the Grow to recovery group delivered by mental health professionals who has received the online training.
  Arms: The Grow to Recovery train-the-trainer group
Other: Control group — Mental health professionals will not receive any training. People with mental illness will receive a spiritual book and read by themselves.
  Arms: Control group

SUMMARY:
Recovery-oriented services are becoming popular in the mental health field. However, recovery-oriented services are still in the beginning stages in Taiwan. Many professionals do not know how to implement recovery-oriented services. More effort should be made to improve mental health services in Taiwan. Hence, the aim of this study is to examine the effectiveness of the Grow to Recovery Train-the-Trainer program.

DETAILED DESCRIPTION:
The study will verify the effectiveness of the Train-the-Trainer program with the cluster randomized controlled trial design. The resesarchers will recruit 10 psychiatric rehabilitation organizations, including 80 mental health professionals and 160 people with mental illness. The professionals of the intervention group will receive a online training and then conduct a 5-month recovery group. The organization-level and service user assessments will be collected to examine the overall outcomes.

ELIGIBILITY:
Inclusion Criteria:

Professionals:

1. working in the community psychiatric rehabilitation organizations
2. being willing to participate in the study

People with mental illness

1. having a diagnosis of mental illness
2. living in the community
3. being age 20 yr or older
4. receiving services from the collaborating organizations
5. filling out the scales independently
6. being able to participate in a recovery group and follow the group rules

Exclusion Criteria:

* attending another recovery-related group

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Recovery Self Assessment (change will be assessed) | Change from Baseline RSA score at 6 months
  The RSA will be used to examine participants' perceptions of the degree to which the organization follows recovery principles. The researchers will collect data from professionals and people with mental illness.
Recovery-Promoting Relationships Scale (change will be assessed) | Change from Baseline RPRS score at 6 months
  The RPRS measures the recovery competence of practitioners from the perspectives of people with mental illness.
Recovery-Promoting Competence Scale (change will be assessed) | Change from Baseline RPCS score at 1.5 month, and 6 months
  The RPCS measures the recovery competence of practitioners and is a self-report scale.
Recovery Attitudes Measure (change will be assessed) | Change from Baseline RAM score at 1.5 month, and 6 months
  The RAM measures the knowledge and attitudes toward recovery.
Stages of Recovery Scale (change will be assessed) | Change from Baseline SRS score at 6 months
  The SRS scale consists of 45 items, with six subscales: the sense of hope, disability management/taking responsibility, regaining autonomy, social functioning/role performance, overall well-being, and willingness to help.
Rosenberg Self-Esteem Scale (change will be assessed) | Change from Baseline RSE score at 6 months
  The purpose of the 10-item RSE scale is to measure self-esteem.
Medical Outcomes Study Social Support Survey (change will be assessed) | Change from Baseline MOS-SS score at 6 months
  The Medical Outcomes Study Social Support Survey (MOS-SS) is a multidimensional, self-administered instrument that addresses all five functions of an interpersonal relationship to assess the various functional dimensions of social support, including emotional , informational, tangible, affectionate, and positive interaction (Sherbourne & Stewart, 1991).
The Hope Scale (change will be assessed) | Change from Baseline THS score at 6 months
  A 12-item THS scale measures level of sense of hope.
Brief Symptom Rating Scale-50 (change will be assessed) | Change from Baseline BSRS-50 score at 6 months
  A BSRS-50 scale comprises 50 items, which best reflect the original ten symptom dimensions and three indices of psychopathology from the SCL-90-R.

OTHER OUTCOMES:
Qualitative data | At 6 month
  The researchers will conduct focus groups with professionals of the intervention group after completing the 5-month recovery group. Those qualitative data will be transcribed and analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No